CLINICAL TRIAL: NCT01950208
Title: The Munich Knee Questionnaire (MKQ) - Development and Validation of a New Patient-reported Outcome Measurement Tool in Knee Surgery
Brief Title: The Munich Knee Questionnaire - Development and Validation
Acronym: MKQ
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Chlodwig Kirchhoff, PD Dr. med., Technical University of Munich
Other Study IDs: Beiromat_01; Kirchhoff_Beiromat (Registry Identifier: Kirchhoff_Beiromat)
Record Dates: First submitted 2013-09-15; First posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Knee Injury
Keywords: Assessment
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- knee pain: patients suffering from knee injury

SUMMARY:
the purpose of this study is to develop and validate a new PRO measurement tool for the knee joint, the so-called Munich Knee Questionnaire (MKQ), allowing for a qualitative self-assessment of the Knee Injury and Osteoarthritis Outcome Score (KOOS), the International Knee Documentation Committee (IKDC), the Lysholm Knee Score, the Western Ontario Meniscal Evaluation Tool (WOMET) and the Tegner Score.

DETAILED DESCRIPTION:
A systematic review of the literature was performed to identify valid and commonly used instruments regarding follow-up examinations in the field of knee surgery. PubMed.gov was searched for knee-specific terms (knee, surgery, joint, lower extremity) combined with psychometric (follow-up, validity, reliability, responsiveness) and instrument-specific terms (self-reported, patient-based, measurement tool, outcome measure, questionnaire). Hence, the KOOS, IKDC, Lysholm, WOMET and Tegner Score were identified as frequent used and valid measurement tools in the evaluation of knee joint function. After analysing each single question of these questionnaires for coincidences regarding measurement of specific knee function, the identified items were condensed to one single question for each specific item. Typical functional abilities (flexion/extension) were depicted as photographs. Thus, one single questionnaire with a total of 33 questions divided in five subscales (Symptoms, Pain, Work and Activities of daily life, Sports and Recreational activities, Physical function and knee related Quality of Life), was created.

ELIGIBILITY:
Inclusion Criteria:

* all patients presenting with knee pain

Exclusion Criteria:

* no exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with knee pain
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Munich Knee Questionnaire (MKQ) | up to 6 weeks starting from onset of symptoms

SECONDARY OUTCOMES:
The self-assessment of the Knee Injury and Osteoarthritis Outcome Score (KOOS) | up to 6 weeks starting from onset of symptoms

OTHER OUTCOMES:
The International Knee Documentation Committee (IKDC) | up to 6 weeks starting from onset of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Chlodwig Kirchhoff, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinik und Poliklinik für Unfallchirurgie, Munich, Bavaria, Germany